CLINICAL TRIAL: NCT00544791
Title: The Effect of Melatonin on Memory and Other Cognitive Function in Patients Diagnosed With Mild Cognitive Impairment (MCI): A Placebo- Controlled Study.
Brief Title: The Effect of Melatonin on Cognitive Function in Patients Diagnosed With Mild Cognitive Impairment
Acronym: MCI
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assaf-Harofeh Medical Center (Other Government)
Collaborators: Neurim Pharmaceuticals Ltd. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 32/07
Record Dates: First submitted 2007-10-14; First posted 2007-10-16 (Estimated); Last update posted 2007-10-16 (Estimated); Status verified 2007-06

CONDITIONS: Mild Cognitive Impairment (MCI)
Keywords: Mild Cognitive Impairment; Melatonin; Antioxidant; Memory; Alzheimer
MeSH Terms: conditions — Cognitive Dysfunction | interventions — Melatonin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Experimental): melatonin 5 mg, daily dose for 6 months
  Interventions: Drug: melatonin
- B (Placebo Comparator)
  Interventions: Drug: placebo like melatonin tablets

INTERVENTIONS:
Drug: melatonin — 5 mg, oral, daily dose for 6 months
  Arms: A
Drug: placebo like melatonin tablets
  Arms: B

SUMMARY:
Recent studies have described the role of melatonin as a sleep regulator and as an anti- oxidative neuroprotective agent in improving sleep quality and delaying cognitive decline in Alzheimer's disease (AD).

In accordance with this data, our hypothesis is that melatonin will delay the cognitive decline in Mild Cognitive Impairment (MCI) patients and reduce the conversion rate from MCI to AD.

ELIGIBILITY:
Inclusion Criteria:

1. MCI assessment according to the Peterson et al. (2001) criteria.
2. Age 55-90 years, inclusive.
3. Study informant available.
4. Mini Mental Status Examination ; MMSE 24-30.
5. Adequate vision and hearing for neuropsychological testing.
6. Normal vitamin B12 level and thyroid function.

Exclusion Criteria:

1. Significant cerebral vascular disease (Modified Hachinski scale > 4).
2. Depression (Hamilton Depression Rating Scale > 12).
3. Central nervous system infarct, infection or focal lesions of clinical significance on CT or MRI scans.
4. Medical diseases or psychiatric disorders that could interfere with study participation.
5. Pregnant, lactating or childbearing potential.
6. Taking vitamin supplements or other supplements.
7. Restrictions on concomitant medication usage, including those with significant cholinergic or anti-cholinergic effects or potential adverse effects on cognition.

Ages: 55 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2007-10; Study Completion 2010-10 (Estimated)

PRIMARY OUTCOMES:
a delay in cognitive decline as measured by memory tests | 6 months

SECONDARY OUTCOMES:
Reduced MCI conversion rate to AD per year | Two years

CONTACTS AND LOCATIONS:
Overall Officials: Micheal khaigrekht, MD, Principal Investigator — Assaf-Harofeh medical center, Memory clinic; Martin Rabey, MD, Principal Investigator — Assaf-Harofeh medical center, Neurology department; Itzhak Sphirer, MD, Study Chair — Assaf-Harofeh medical center, sleep lab; Ran Shorer, MA, Study Chair — Asaf Harofeh medical center, Memory clinic
Locations (1):
- Memory clinic, 'Asaf Harofeh' medical center, Ẕerifin, Israel